CLINICAL TRIAL: NCT02710084
Title: Piloting Treatment With Intranasal Oxytocin in Phelan-McDermid Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander Kolevzon (Other)
Responsible Party: Sponsor-Investigator, Alexander Kolevzon, Alexander Kolevzon, Clinical Director, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 15-1223
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Phelan-McDermid Syndrome
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): The first phase of the study will follow a double-blind, placebo-controlled design. Participants randomized to the experimental group will receive intranasal oxytocin in doses of 24 IU, two times daily, for a total of 48 IU. Doses may be reduced by 8 IU/day if safety concerns emerge. During the second phase of the study, all participants will receive oxytocin, in identical doses.
  Interventions: Drug: Oxytocin
- Saline (Placebo Comparator): During the first phase, patients randomized to the placebo group will receive intranasal saline solution in doses of 24 IU two times daily, for a total of 48 IU. During the second phase of the study, all participants will receive oxytocin, in identical doses.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — Intranasal oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Saline — Placebo
  Arms: Saline

SUMMARY:
This is a pilot study examining the efficacy, safety and tolerability of intranasal oxytocin as a novel treatment in Phelan-McDermid syndrome (PMS). This study will utilize a randomized, placebo-controlled design for 12 weeks (phase 1), followed by an open-label extension for 12 weeks (phase 2). The purpose is to evaluate the effect of intranasal oxytocin on impairments in attention, social memory, socialization, language, and repetitive behaviors.

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of Phelan-McDermid syndrome defined by pathogenic deletion or mutation of the SHANK3 gene and confirmed by chromosomal microarray or sequencing.
* Must be between the ages of 5 and 17
* Must be on stable medication and psychosocial therapy regimens for at least three months prior to enrollment

Exclusion criteria:

* Allergy to oxytocin
* Active cardiovascular disease, epilepsy, or renal disease that is not controlled by medication
* Pregnant, lactating or refuse to practice contraception if sexually active
* Have caretakers who are unable to speak English, be consistently present at visits to report on symptoms, or are otherwise judged unable to comply with the protocol by the study team
* Comorbid conditions such that the patient is too medically compromised to participate

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-04-29; Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fastman J, Foss-Feig J, Frank Y, Halpern D, Harony-Nicolas H, Layton C, Sandin S, Siper P, Tang L, Trelles P, Zweifach J, Buxbaum JD, Kolevzon A. A randomized controlled trial of intranasal oxytocin in Phelan-McDermid syndrome. Mol Autism. 2021 Sep 30;12(1):62. doi: 10.1186/s13229-021-00459-1. PMID 34593045

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Then Oxytocin: During the first phase, patients randomized to the placebo group received intranasal saline solution in doses of 24 IU two times daily, for a total of 48 IU. During the second phase of the study, all participants received intranasal oxytocin, in identical doses.
- Intranasal Oxytocin: The first phase of the study followed a double-blind, placebo-controlled design. Participants randomized to the experimental group received intranasal oxytocin started the trial with a dose of 24 international units (IU) twice daily (BID), which was adjusted to 12 IU BID, subsequently the dose was increased to 24IU BID. Each insufflation delivered 4 IU and three insufflations (12 IU) in each nostril were given twice daily for a total daily dose of 48 IU. The second phase was a 12-week open-label extension phase during which all participants received intranasal oxytocin.
Period: First Phase - 12 Weeks
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Started | 10 | 8
Completed | 7 | 7
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: Open Label Phase: Week 12 to 24
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (3.6) | 6.8 (1.4) | 8.4 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Aberrant Behavior Checklist Social Withdrawal (ABC-SW) subscale [Mean (Standard Deviation); unit: units on a scale] — 16 items, Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). Total scores range from 0 to 48, with higher scores indicating poorer health outcomes.
  units on a scale | 20.1 (6.1) | 14. (3.4) | 17.4 (5.9)
Verbal DQ - developmental quotient [Mean (Standard Deviation); unit: T-score] — Developmental quotients are calculated by averaging the age equivalent (AE) scores of the components, dividing by chronological age, and multiplying by 100. The verbal DQ (VDQ) includes Expressive Language (EL) and Receptive Language (RL). The average (mean) is 100 with a standard deviation of 15 points. Higher scores indicate greater cognitive ability.
  T-score | 14.9 (12.8) | 26.4 (21.3) | 20 (17.6)
Nonverbal DQ [Mean (Standard Deviation); unit: T-score] — Developmental quotients are calculated by averaging the age equivalent (AE) scores of the components, dividing by chronological age, and multiplying by 100. The nonverbal DQ (NVDQ) includes scales of Visual Reception (VR) and Fine Motor (FM) abilities. The average (mean) is 100 with a standard deviation of 15 points. Higher scores indicate greater cognitive ability.
  T-score | 20.1 (11.7) | 26.1 (13.1) | 22.7 (12.3)
Full Scale DQ [Mean (Standard Deviation); unit: T-score] — Developmental quotients are calculated by averaging the age equivalent (AE) scores of the components, dividing by chronological age, and multiplying by 100. The average (mean) is 100 with a standard deviation of 15 points. Higher scores indicate greater cognitive ability. An IQ below 70 is part of the diagnostic criteria for intellectual disability.
  T-score | 17.4 (11.8) | 26.3 (16.7) | 21.4 (14.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Aberrant Behavior Checklist
Description: Change in scale at week 12 as compared to baseline. Aberrant Behavior Checklist - behavior rating subscales for the assessment of treatment effects.16 items, Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). Total score range from 0 to 48, with higher score indicating poorer health outcomes.
Time Frame: Baseline and Week 12
Population: In the case of two participants who dropped out after week 4, difference scores were calculated for each outcome measure using the last observation carried forward (This is why some measures have N's of 9 and 7). Two participants dropped out after BL and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 9 | 7
score on a scale
  Social Withdrawal | -7.44 (4.58) | -2.42 (3.15)
  Irritability | -5 (6.63) | -1.71 (7.13)
  Stereotypy | -2.22 (4.66) | 0.57 (2.99)
  Hyperactivity | -8.11 (11.85) | -2.71 (7.34)
  Inappropriate speech | -1.67 (3.04) | -7.14 (2.21)

2. Secondary Outcome: Change in Visual Paired Comparison (VPC) Task
Description: Change in VPC Task has 2 subscores at week 12 as compared to baseline. The subject is initially presented with a target for familiarization and the familiar target is then paired with a novel target. Recognition is indexed by a novelty score derived from the percentage of time looking at the novel stimulus vs. the familiar stimulus. The Social-Novel Preference score refers to the proportion of time spent looking at novel stimuli out of all the time spent looking at both novel and familiar stimuli in the social test. The Nonsocial-Novel Preference score refers to the proportion of time spent looking at novel stimuli out of all the time spent looking at both novel and familiar stimuli in the nonsocial test.The scores are given in proportions with a range from -1 to 1. A score of -1 would mean the participant shows a preference for familiar stimuli and a score of 1 demonstrates a preference for novel stimuli.
Time Frame: Baseline and Week 12
Population: Only 3 participants with data from baseline and week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 1 | 2
score on a scale
  Social-Novel Preference | 0.01 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated. | 0.02 (0.12)
  Nonsocial-Novel Preference | -0.38 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated. | 0.22 (0.12)

3. Secondary Outcome: Change in Gap-Overlap Task
Description: One of three computerized eye tracking tasks to measure attention. three computer screens are set up side by side. A stimulus initially appears on the central screen, and once the participant orients to that stimulus, another stimulus will appear on one of the lateral screens. In the "gap" condition, the central stimulus will disappear before the peripheral stimulus appears. In the "overlap" condition, the central stimulus will remain on the screen while the peripheral stimulus appears. In both conditions, reaction times of the participant's eye movements (saccadic reaction time) from the central stimulus to the peripheral stimulus will be measured. Gap Effect measures the difference between average Gap and Overlap saccade latencies.
Time Frame: Baseline and Week 12
Population: Only 2 participants with data from both baseline and Week 12
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 2 | 0
milliseconds (ms) | 63.81 (34.19) |

4. Secondary Outcome: Change in Flicker Tasks
Description: One of three computerized eye tracking tasks to measure attention. The "flicker task," or the four-alternative forced-choice preferential looking paradigm - the time interval over which the visual system is able to parse information. Scores range from -1 to 1 with higher scores indicating better (more typical) performance.
Time Frame: Baseline and Week 12
Population: Only 1 participant with data from baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 0 | 1
score on a scale
  Preference for the Target Box at 0.2 Hz |  | 0.10 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated.
  Preference for the Target Box at 0.5 Hz |  | 0.30 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated.
  Preference for the Target Box at 1 Hz |  | -0.12 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated.
  Preference for the Target Box at 2 Hz |  | 0.03 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated.

5. Secondary Outcome: Change in Vineland Adaptive Behavior Scales
Description: Mean change in scale at week 12 as compared to baseline. Vineland Adaptive Behavior Communication Domain measures adaptive functioning.
  Vineland-II subdomains (Communication, Daily Living Skills, Socialization, Motor, Adaptive Behavior Composite, Internalizing, Externalizing and maladaptive) are V-scale scores (M=15, SD=3). Higher scores indicate better developed adaptive social behavior.
  Vineland-II domain and composite values are standard scores (M=100, SD=15). Higher scores indicate better developed adaptive social behavior.
Time Frame: Baseline and Week 12
Population: Participants were only included in this analysis if they had Vinelands at BL and Week 12. One incomplete Maladaptive subdomain form for one participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 7 | 6
score on a scale
  Communication | 4 (7.72) | 2.83 (4.83)
  Daily Living Skills | 3.29 (8.39) | 1.17 (5.13)
  Socialization | 3 (4.86) | -0.5 (4.46)
  Motor: number analyzed (Participants) | 6 | 6
  Motor | 1 (3.46) | 3.17 (6.18)
  Adaptive Behavior Composite | 3.14 (3.80) | 2 (3.22)
  Internalizing | -1.14 (1.07) | 6 (0.84)
  Externalizing | -1.14 (2.73) | 6 (1.33)
  Maladaptive: number analyzed (Participants) | 6 | 6
  Maladaptive | -1.33 (2.42) | 6 (0.55)

6. Secondary Outcome: Change in Repetitive Behavior Scale-Revised (RBS-R)
Description: Change in Repetitive Behavior Scale at week 12 as compared to baseline. the RBS-R is a 44-item self-report questionnaire consisting of subscales and one additional global rating score from 1-100. Score range for Stereotypic Behavior subscale is 0-27, Self-Injurious Behavior subscale is 0-24, Compulsive Behavior subscale is 0-18, Ritualistic/Sameness Behavior subscale is 0-36, and Restricted Interests subscale 0-9. Total scale for RBS-R is 0-214, with higher score indicating more severe problem.
Time Frame: Baseline and Week 12
Population: Patients were only included in this analysis if they had RBS-R at BL and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 9 | 7
score on a scale
  Stereotypic behaviors | -1.67 (2.78) | 0.29 (2.87)
  Self-injury | -1.22 (3.11) | 1 (2.31)
  Compulsive behaviors | -1.56 (3.09) | -0.14 (0.69)
  Ritualistic behaviors | -1.33 (2.40) | -0.43 (1.62)
  Sameness behaviors | -2 (2.65) | -0.29 (1.60)
  Restrictive behaviors | -1.43 (2.39) | 0.14 (0.90)
  Overall Score | -8.56 (13.29) | 0 (5.56)

7. Secondary Outcome: Change in Clinical Global Impression - Severity Scales
Description: Mean Change in Clinical Global Impression-Severity Scales at week 12 as compared to baseline. Clinical Global Impressions (CGI) Rating Scales are commonly used to measure symptom severity and global improvement in treatment studies of patients with developmental disorders. There Severity Scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of illness at the time of assessment. Full scale from 1 - 7. Higher scores indicate greater symptom severity.
Time Frame: Baseline and Week 12
Population: Data from all participants who had data collected at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 9 | 7
score on a scale | -0.11 (0.17) | -0.1 (0.24)

8. Secondary Outcome: Change in Short Sensory Profile (SSP)
Description: Mean Change in Short Sensory Profile Scale at week 12 as compared to baseline, measuring sensory sensitivity and sensory seeking behavior. The SSP is a 38-item caregiver questionnaire. Items are based on a 5-point Liker scale ranging from 1=always to 5=never. Tactile Sensitivity ranges from 7-35. Taste/Smell Sensitivity ranges from 4-20. Movement Sensitivity ranges from 3-15. Underresponsive/Seeks Sensation ranges from 7-35. Auditory Filtering ranges from 6-30. Low Energy/Weak ranges from 6-30. Visual/Auditory Sensitivity ranges from 5-25. Total scale range from 38-190. Lower scores indicate a higher probability of sensory processing abnormalities.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 9 | 7
score on a scale
  Tactile | 2.56 (5.17) | 1.57 (3.78)
  Taste/Smell | 1.67 (2.88) | 0.71 (1.89)
  Movement | -0.67 (2.0) | 0.29 (0.76)
  Under-responsive/seeks attention | 4.44 (5.50) | 0.71 (4.68)
  Auditory filtering | 4 (5.68) | 0.29 (5.21)
  Low energy/weak | 1.67 (6.18) | -0.71 (4.19)
  Visual/auditory sensitivity | 1.89 (2.57) | -0.86 (2.67)
  Summary total | 14.33 (21.31) | 1 (17.95)

9. Secondary Outcome: Change in Macarthur-Bates Communicative Development Inventory (MCDI)
Description: Macarthur-Bates Communicative Development Inventory at week 12 as compared to baseline, measuring language. Words and Gestures Forms are for children ages 8-18 months. In the form, the first part prompts parents to document the child's understanding of hundreds of early vocabulary items separated into semantic categories such as animal names, household items, and action words. Parents mark the words understood or used, and the forms yield separate indexes of words understood and words produced. The second part of each form asks parents to record the communicative and symbolic gestures the child has tried or completed. Ranges for each subscale score are as follows: Phrases understood (0-28), Words understood (0-396), Words produced (0-396), Early gestures (0-18), Later gestures (0-45), Total gestures (0-63). Higher scores indicate a great number of words, phrases, or gestures understood or produced.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 7 | 7
score on a scale
  Phrases understood | 0.83 (6.62) | 1.43 (3.55)
  Words understood | -9.17 (52.59) | 7 (13.41)
  Words produced | 11.67 (41.90) | 2.57 (10.23)
  Early gestures | 1.83 (2.64) | 0.29 (1.38)
  Later gestures | 3 (7.48) | 0.86 (1.95)
  Total gestures | 4.83 (9.97) | 0.57 (2.07)

10. Secondary Outcome: Change in EEG Tasks: Auditory Habituation
Description: In the Auditory Habituation EEG task, participants listen to a series of 4 tones and the neural responses to each of these tones (event related potentials, ERPs ) are averaged. The N1 and P2 components are typical responses to auditory stimuli. The N1 response is the initial, quick response to hearing a stimulus, and P2 reflects the later processing of the stimulus. Both of these should be greater in response to the first tone, and then reduce in response to each subsequent tone. This is known as habituation, and is calculated as the change in Tone 1 minus Tone 2 response for both N1 and P2 components.
Time Frame: Baseline and Week 12
Population: Data results available only for those who underwent Auditory Habituation EEG task
Measure: Mean (Standard Deviation); unit: microvolts (µV)
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 2 | 1
microvolts (µV)
  Auditory Habituation: N1 Habituation Change | 0.05 (0.37) | 0.12 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated.
  Auditory Habituation: P2 Habituation Change | 1.15 (0.91) | -3.48 (NA) — Data collected from 1 participant and hence the measure of dispersion (i.e., standard deviation) cannot be calculated.

11. Secondary Outcome: Number of Adverse Events
Description: Number of Adverse Events through week 12
Time Frame: week 12
Measure: Number; unit: events
Groups:
- Intranasal Oxytocin: The first phase of the study will follow a double-blind, placebo-controlled design. Participants randomized to the experimental group will receive intranasal oxytocin started the trial with a dose of 24 international units (IU) twice daily (BID), which was adjusted to 12 IU BID, subsequently the dose was increased to 24IU BID. Each insufflation delivered 4 IU and three insufflations (12 IU) in each nostril were given twice daily for a total daily dose of 48 IU.
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 10 | 8
events | 41 | 35

12. Secondary Outcome: Change in Caregiver Strain Index
Description: Mean Change Caregiver Strain Index at week 12 as compared to baseline. The Caregiver Strain Questionnaire is a 21-item measure of self-reported strain experienced by caregivers and families of youth with emotional problems, with responses on a 5-point Likert scale (0 = Not at all, 4 = very much). Full scale from 0 to 84, higher score indicates higher caregiver burden
Time Frame: Baseline and Week 12
Population: incomplete form for one participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 6 | 7
score on a scale | -1.83 (1.47) | -0.86 (1.07)

13. Secondary Outcome: Change in Mullen Scales of Early Learning (MSEL)
Description: Change in Mullen Scales of Early Learning (MSEL) at week 12 as compared to baseline. The Mullen Scales results are reported using Age Equivalents, which provides an estimate of the chronological age (CA) in years and months at which a typically developing child demonstrates the skills displayed by the child being assessed. The Mullen Scales results are reported using T scores. (M = 100, SD = 15). Each subscale is standardized to calculate an age-equivalent score. Higher scores represent a higher CA, and therefore better outcome.
Time Frame: baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Saline Then Oxytocin | Intranasal Oxytocin
Number analyzed (Participants) | 7 | 7
T-score
  Gross motor | -1.57 (4.69) | -0.86 (1.46)
  Visual Reception | 0.29 (7.0) | 2.86 (3.30)
  Fine Motor | -0.29 (1.11) | 0.71 (1.80)
  Receptive Language | -1.86 (4.86) | 1.71 (2.70)
  Expressive Language | 0.43 (2.61) | 0.43 (1.80)

ADVERSE EVENTS:
Time Frame: through week 12
Description: Monitoring of adverse events (AEs) was done using an adapted semi-structured interview, the Safety and Monitoring Uniform Report Form (SMURF). AEs were documented with respect to severity, duration, management, relationship to study drug, and outcome. Severity was graded using a scale of mild, moderate, or severe.
Groups:
- Saline: During the first phase, patients randomized to the placebo group received intranasal saline solution in doses of 24 IU two times daily, for a total of 48 IU.
- Intranasal Oxytocin: The first phase of the study followed a double-blind, placebo-controlled design. Participants randomized to the experimental group received intranasal oxytocin started the trial with a dose of 24 international units (IU) twice daily (BID), which was adjusted to 12 IU BID, subsequently the dose was increased to 24IU BID. Each insufflation delivered 4 IU and three insufflations (12 IU) in each nostril were given twice daily for a total daily dose of 48 IU. During the second phase of the study, all participants received oxytocin, in identical doses.
Arm/Group | Saline | Intranasal Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/10 | 15/15
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/15
Other Adverse Events (participants affected / at risk) | 9/10 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline (N=10) | Intranasal Oxytocin (N=15)
Sedation (General disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Periorbital / facial swelling (General disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Sleep disturbance (General disorders) | 2 | 7
Increased appetite (Metabolism and nutrition disorders) | 1 | 1
Irritability/agitation (Psychiatric disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Runny nose/congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fever (General disorders) | 4 | 9
Aggression/self-injury (Psychiatric disorders) | 1 | 2
Infection (Infections and infestations) | 3 | 6
Elated mood/Silliness (Psychiatric disorders) | 1 | 5
Leg weakness (General disorders) | 1 | 1
Restlessness/hyperactivity (Psychiatric disorders) | 1 | 8
Bloody nose (General disorders) | 0 | 3
Stereotypies (Psychiatric disorders) | 2 | 4
Apathy (Psychiatric disorders) | 0 | 1
Foot pain (General disorders) | 1 | 0
Hirsutism (Endocrine disorders) | 0 | 1
Tooth pain (Gastrointestinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3
Allergies/asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Enuresis (Renal and urinary disorders) | 1 | 1
Accidental injury (Injury, poisoning and procedural complications) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Rubbing ears (Ear and labyrinth disorders) | 1 | 0
Disinhibited (Psychiatric disorders) | 1 | 1
Oppositional behavior (Psychiatric disorders) | 3 | 2
Low frustration tolerance (Psychiatric disorders) | 1 | 3
Tantrums (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The small sample size, potential challenges with drug administration, and expectancy bias due to relying on parent reported outcome measures may all contribute to limitations in interpreting results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT02710084/Prot_SAP_000.pdf